CLINICAL TRIAL: NCT04642118
Title: Low-pressure Pulmonary Recruitment Maneuver to Decrease Post-laparoscopic Shoulder Pain in Gynecologic Surgery: A Double-blind Randomized Placebo Controlled Trial
Brief Title: Low-pressure Pulmonary Recruitment Maneuver to Decrease Post-laparoscopic Shoulder Pain in Gynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 147/2563
Record Dates: First submitted 2020-08-28; First posted 2020-11-24 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2020-08

CONDITIONS: Gynecologic Disease; Laparoscopic Surgery
Keywords: Low pressure; Pulmonary Recruitment Maneuver; Post-laparoscopic Shoulder Pain
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pulmonary recruitment maneuver 30 cmH2O (Experimental): After laparoscopic surgery has finished in operator room (before moving off trocar), patient will be set in Trenderlenberg position (Tilted head low) and then surgeon will compress abdomen to release residual gas after operation about 2 minutes.
  The patients in this group will be received positive pressure from Pulmonary recruiment maneuver [balloon bag] from anesthesiologist 5 times of setting pressure 30 cmH2O, 5 seconds per time to increase indirect abdominal pressure to release residual gas
  Interventions: Procedure: Pulmonary recruitment maneuver
- Pulmonary recruitment maneuver 40 cmH2O (Active Comparator): After laparoscopic surgery has finished in operator room (before moving off trocar), patient will be set in Trenderlenberg position (Tilted head low) and then surgeon will compress abdomen to release residual gas after operation about 2 minutes.
  The patients in this group will be received positive pressure from Pulmonary recruiment maneuver [balloon bag] from anesthesiologist 5 times of setting pressure 40 cmH2O, 5 seconds per time to increase indirect abdominal pressure to release residual gas
  Interventions: Procedure: Pulmonary recruitment maneuver
- Control (No Intervention): After laparoscopic surgery has finished in operator room (before moving off trocar), patient will be set in Trenderlenberg position (Tilted head low) and then surgeon will compress abdomen to release residual gas after operation about 2 minutes.
  The patients in this group will not be received any positive pressure from Pulmonary recruiment maneuver [balloon bag] from anesthesiologist.

INTERVENTIONS:
Procedure: Pulmonary recruitment maneuver — Using setting pressure form ventilator to increase pulmonary pressure by compress balloon bag 5 times, 5 seconds per time
  Arms: Pulmonary recruitment maneuver 30 cmH2O; Pulmonary recruitment maneuver 40 cmH2O

SUMMARY:
Research objective to compare outcomes (shoulder pain score, wound pain score, post-operative residual pneumoperitoneum, lung complication, GI discomfort, administered additional analgesics, time to hospital staying) of using Pulmonary Recruitment maneuver with pressure 30 cmH2O, 40 cm H2O and control group in women with post laparoscopic gynecologic surgery in Rajavithi hospital.

DETAILED DESCRIPTION:
Research design is Randomized control trial. The women who go to laparoscopic gynecologic surgery don't know the allocation. Women will be randomizes in to 3 group: PRM 30 cmH2O, 40 cmH2O and control

After laparoscopic surgery has finished in operator room (before moving off trocar), woman all group will be set in Trenderlenberg position (Tilted head low) and then surgeon will compress abdomen to release residual gas after operation about 2 minutes.

The patients in group of using Pulmonary Recruitment Maneuver will be received positive pressure from balloon bag from anesthesiologist 5 times of setting pressure [30 cmH2O, 40 cmH2O], 5 seconds per time to increase indirect abdominal pressure to release residual gas

After surgery at 12, 24 and 48 hours, patients will be follow up and evaluate shoulder and wound pain. Chest X-ray will be done to evaluate residual pneumoperitoneum and lung complication. GI discomfort, administered additional analgesics and time to hospital staying will be evaluated and recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Anesthesiologists physical status (ASAPS) classification I-II
* Absence of Pregnancy
* With inform-consent

Exclusion Criteria:

* Inability to accurately express pain
* Past history of shoulder or lung surgery
* Chronic shoulder problem
* Epigastric pain
* Lung disease such as emphysema or pneumothorax
* Severe kidney or liver disease
* Drug allergy (NSAIDs, Paracetamol)
* On current medication: corticosteroid
* Psychiatric disorder

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
shoulder pain from using PRM 30 cmH2O | During stay in hospital around 2-3 days
  To compare shoulder pain score(Visual analogue scale from score 0(no pain) to score 10 (maximum pain)) after laparoscopic gynecologic surgery between PRM at 30 cmH2O group and control group at 12, 24 and 48 hrs.

SECONDARY OUTCOMES:
wound pain | During stay in hospital around 2-3 days
  evaluate with Visual analogue scale from score 0(no pain) to score 10 (maximum pain)
shoulder pain from using PRM 40 cmH2O | During stay in hospital around 2-3 days
  To compare shoulder pain score(Visual analogue scale from score 0(no pain) to score 10 (maximum pain)) after laparoscopic gynecologic surgery between PRM at 40 cmH2O group and control group at 12, 24 and 48 hrs.
Post-operative residue pneumoperitoneum | after surgery in day 1
  Residue air volume in abdominal cavity will be measured (Hight from diaphragm to upper border of liver (cm.)) from Chest x-ray PA upright
Lung complication | after surgery in day 1
  Number of participants with complication (incident) such as pneumothorax, Lung atelectasis, Pleural effusion etc. will be recorded
GI discomfort | during stay in hospital around 2-3 days
  number of symptom
Time to hospital staying | During stay in hospital around 2-3 days
  record day which stay in hospital with abnormal condition
Administered additional analgesics | During stay in hospital around 2-3 days
  number of morphine using

CONTACTS AND LOCATIONS:
Overall Officials: Anon Yodruangwong, Study Director — Resident
Locations (1):
- Rajavithi hospital, Bangkok, Thailand